CLINICAL TRIAL: NCT05759234
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of HS248 in the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Study of HS248 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanhui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS248-I-01
Record Dates: First submitted 2023-02-07; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: At this stage, it is planned that HS248 will adopt the traditional "3+3" method of increasing doses at four dose levels of 20 mg, 40 mg, 60 mg and 80 mg. All dosage components are divided into single administration stage and multiple administration stage. After 5 days of observation after single administration, it enters the stage of multiple administration. In the stage of multiple administration, HS248 is administered once a day (qd) for 28 days. a treatment cycle. 33 days after the first administration (the 5-day observation period in the single-administration phase and the first cycle in the multiple-administration phase) is the dose-limiting toxicity (DLT) observation period of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS248 pieces (Experimental): dose escalation period： At this stage, it is planned that HS248 will adopt the traditional "3+3" method of increasing doses at four dose levels of 20 mg, 40 mg, 60 mg and 80 mg. All dosage components are divided into single administration stage and multiple administration stage. After 5 days of observation after single administration, it enters the stage of multiple administration. In the stage of multiple administration, HS248 is administered once a day (qd) for 28 days. a treatment cycle. 33 days after the first administration (the 5-day observation period in the single-administration phase and the first cycle in the multiple-administration phase) is the dose-limiting toxicity (DLT) observation period of this study
  Interventions: Drug: HS248 pieces

INTERVENTIONS:
Drug: HS248 pieces — The overall safety and tolerability of PI3Kγ inhibitor monotherapy for solid tumors is good, and it has shown preliminary clinical benefits. The safety of PI3Kγ inhibitor combined with immune checkpoint inhibitor is good, and the efficacy of single drug is significantly improved. Based on the evaluation of the safety and efficacy results of HS248 preclinical and clinical studies of similar PI3Kγ inhibitors, the benefits of this product outweigh the risks for patients with advanced solid tumors who have progressed through standard treatment, have toxicity intolerance, or have no standard treatment regimen. Sufficient to support planned clinical studies.

SUMMARY:
This study is a non-random, open multi-center study This study is a non-random, open multi-center phase I study, aimed at evaluation period research, aimed at In the evaluation phase study, it aims to evaluate the safety, tolerance PK characteristics and preliminary anti-tumor activity of HS248 in patients with advanced solid tumors. The study was divided into 2 phases, including dose escalation and dose expansion。

DETAILED DESCRIPTION:
Main purpose:

Assess the safety and tolerability of HS248 in patients with advanced solid tumors, and determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of HS248.

Secondary purpose: Secondary purpose:

Assess the pharmacokinetic (PK) profile of HS248 in patients with advanced solid tumors; To evaluate the preliminary antitumor activity of HS248 in patients with advanced solid tumors. Preliminary antitumor activity in patients with advanced solid tumors.

Other purposes:

Population-based PK (PopPK) analysis method, exploratory description) analysis method, exploratory description) analysis method, exploratory description) analysis method, exploratory description of HS248 in patients with advanced solid tumors PK features in; Evaluate the relationship between exposure and efficacy and adverse events (AEs) of HS248 in patients with advanced solid tumors, as data permit; To explore the changes of HS248 in myeloid-derived suppressor cells (MDSC) and CD8+ T cells in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical trial, understand and follow the research procedures and voluntarily sign the ICF;
2. Male or female, age ≥18 when signing the ICF;
3. Expected survival period ≥ 12 weeks;
4. Patients with advanced solid tumors confirmed by histology/cytology, who have progressed through standard treatment, have toxicity intolerance, or have no standard treatment plan (patients with multiple solid tumors are included in the dose-escalation phase, and the population included in the dose-expansion phase will be based on dose escalation phase study data and the potential advantageous population of similar drugs);
5. Eastern Cooperative Oncology Group (ECOG) physical status score 0-1

Exclusion Criteria:

1. Symptomatic or untreated central nervous system metastasis or primary central nervous system malignancy;
2. Other known malignant tumors in the past 5 years, except cured localized tumors, including carcinoma in situ of the cervix, basal cell carcinoma of the skin, and carcinoma in situ of the prostate;
3. Previous history of autoimmune diseases, stem cell transplantation or organ transplantation;
4. Known drug-induced liver injury, chronic active hepatitis, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, persistent extrahepatic obstruction caused by gallstones, cirrhosis or portal hypertension;
5. Peptic ulcer and/or gastrointestinal bleeding at present or in the past;
6. Gastrointestinal dysfunction that may limit the absorption of the test drug, including motility disorders, malabsorption syndrome or inflammatory bowel disease;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From first dose of HS248 through 28 days after the last HS248 treatment (up to 2 years); each cycle is 28 days
  To examine the incidence of clinical and laboratory adverse events after multiple doses of HS-248 in the dose escalation and dose expansion phases
MTD and/or RP2DP2D | The end of the study is defined as the last subject completing the last visit, study treatment for 2 years, loss to follow-up, death or withdrawal of informed consent, whichever occurs first
  MTD and/or RP2DP2D

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | From date of initial dose until up to 33 days for treatment
  Cmax of HS248
Area Under the Plasma Concentration versus Time Curve (AUC) | From date of initial dose until up to 33 days for treatment
  AUC of HS248
ORR | Up to 2 years
  Objective Response Rate
DOR | Up to 2 years
  Duration of Remission
PFS | Up to 2 years
  Progression-Free Survival
DCR | Up to 2 years
  Disease Control Rate
OS | Up to 2 years
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No